CLINICAL TRIAL: NCT07139652
Title: Patient and Clinician Perceptions of Safe Ambulation and Their Association With Clinical Outcomes in Individuals With Incomplete Spinal Cord Injury: An Observational Study
Brief Title: Patient and Clinician Perceptions of Safe Ambulation in Incomplete Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: AnkaraCHBilkent-PMR-MSS-05
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injuries (SCI)
Keywords: Spinal Cord Injury; Walking; Rehabilitation; Self Report; Perception
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with Incomplete Spinal Cord Injury: Adults (≥18 years) with incomplete spinal cord injury (ASIA C or D) at T3 or lower levels, admitted to an inpatient rehabilitation program. All participants undergo standardized clinical and questionnaire-based assessments, including the Walking Index for Spinal Cord Injury II (WISCI II), patient-rated and therapist-rated ambulation levels, lower extremity muscle strength, gait speed, balance, functional independence, and quality of life. Fall history and assistive device preferences are also recorded. No control group is included.

SUMMARY:
This observational cross-sectional study aims to investigate the relationship between patient and therapist perceptions of safe ambulation and objective clinical outcomes in individuals with incomplete spinal cord injury (iSCI). Adults with iSCI at T3 or lower levels (ASIA C or D) admitted to an inpatient rehabilitation program are assessed for walking status using the Walking Index for Spinal Cord Injury II (WISCI II), including patient-rated and therapist-rated levels. Secondary outcomes include lower extremity muscle strength, gait speed, timed up and go, balance, functional independence, quality of life, fall risk, and assistive device preferences. The study seeks to identify the extent to which patient and therapist perceptions align with objective measures and to explore their associations with fall history and functional outcomes, aiming to improve discharge planning and fall prevention strategies.

DETAILED DESCRIPTION:
This observational, cross-sectional study was conducted to examine the relationship between perceived and actual safe ambulation levels in individuals with incomplete spinal cord injury (iSCI) and their association with key clinical outcomes. Adult participants (≥18 years) with traumatic or non-traumatic iSCI at T3 or lower levels (ASIA C or D) admitted to an inpatient rehabilitation program were included. Exclusion criteria were inability to provide informed consent or severe cognitive impairment (Mini-Mental State Examination score < 25).

The primary outcome was walking status, assessed using the Walking Index for Spinal Cord Injury II (WISCI II). Both patient-rated (P13) and therapist-rated (T5) WISCI II levels were recorded to capture perceived safe ambulation limits. Secondary outcomes included lower extremity muscle strength (LEMS), 10-Meter Walk Test (10MWT), Timed Up and Go (TUG), Berg Balance Scale (BBS), Spinal Cord Independence Measure III (SCIM III), and WHOQOL-BREF-TR for health-related quality of life. Additional questionnaires assessed fall risk perception, assistive device preferences, readiness for discharge, coping strategies, acceptance and action levels, and assistive technology satisfaction.

Gait parameters were measured on a C-Mill® treadmill platform, including step time, stance phase percentage, stride length, step width, cadence, gait speed, and double support time. Falls and near-fall incidents in the past year were self-reported. Data were analyzed to determine correlations between perception-based and performance-based measures and to explore the relationship between discrepancies in patient and therapist ratings with fall frequency and functional independence.

The study aims to provide evidence to guide clinical decision-making in rehabilitation, optimize discharge planning, reduce fall risk, and improve the integration of patient perspectives into therapy planning for individuals with iSCI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of incomplete spinal cord injury (ASIA C or D) at T3 or lower neurological level

Exclusion Criteria:

* Refusal to participate
* Communication impairment severe enough to prevent obtaining information from the participant (e.g., mental problems, confusion, coma)
* Mini-Mental State Examination score < 25

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) with incomplete spinal cord injury (ASIA C or D) at T3 or lower neurological level, admitted to a rehabilitation program. Participants present a range of functional ambulation abilities and use various assistive devices. Both male and female patients with traumatic or non-traumatic etiology are included.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Walking Index in Spinal Cord Injury II | Baseline (single time point, within 24-month recruitment period)
  Walking Index for Spinal Cord Injury II (WISCI II), which assessed walking independence and the need for assistive devices. Scores ranged from 0 to 20 based on the amount of physical assistance, use of braces, and walking aids required to walk 10 meters. In addition to the measured WISCI II score, patient-rated WISCI II (P13) and therapist-rated WISCI II (T5) levels were recorded to reflect the levels at which the individual and the clinician perceived safe ambulation.

SECONDARY OUTCOMES:
ASIA Lower Extremity Muscle Score | Baseline (single time point, within 24-month recruitment period)
  Assessment of lower extremity muscle strength using the American Spinal Injury Association (ASIA) Lower Extremity Motor Score (LEMS)
Ten-Meter Walking Test | Baseline (single time point, within 24-month recruitment period)
  Ten-Meter Walking Test for overground walking speed assessment
Timed Up and Go Test | Baseline (single time point, within 24-month recruitment period)
  Timed Up and Go Test overground walking assessment
Berg Balance Scale | Baseline (single time point, within 24-month recruitment period)
  Berg Balance Scale for balance assessment
Spinal Cord Independence Measure (SCIM III) | Baseline (single time point, within 24-month recruitment period)
  Spinal Cord Independence Measure (SCIM III) for activity of daily living assessment
World Health Organization Quality of Life Scale-Short Form (WHOQOL - BREF) | Baseline (single time point, within 24-month recruitment period)
  World Health Organization Quality of Life Scale-Short Form (WHOQOL - BREF) for quality of life assessment
Quebec User Evaluation of Satisfaction with Assistive Technology 2.0 (QUEST 2.0) | Baseline (single time point, within 24-month recruitment period)
  A questionnaire evaluating user satisfaction with assistive devices in terms of performance and service quality.
RHDS/SF | Baseline (single time point, within 24-month recruitment period)
  The RHDS/SF assessed patients' self-perceived readiness for hospital discharge and ability to manage care needs at home, with scores from 0 to 10 where higher scores indicated greater readiness.
Acceptance and Action Questionnaire - II (AAQ-II) | Baseline (single time point, within 24-month recruitment period)
  The AAQ-II measured psychological flexibility and experiential avoidance using nine items rated from 1 (never true) to 7 (always true), with lower scores indicating greater flexibility.
Spinal Cord Lesion-Related Coping Strategies Questionnaire (SCLCSQ) | Baseline (single time point, within 24-month recruitment period)
  The SCLCSQ assessed coping strategies in individuals with spinal cord injury across three domains-acceptance, social confidence, and fighting spirit-using 12 items rated on a 4-point scale.
P1 - Fear of falling during daily ambulation with preferred assistive device/orthosis (Visual Analog Scale) | Baseline (single time point, within 24-month recruitment period)
  P1 assessed the patient's fear of falling during daily ambulation with their preferred assistive device or orthosis on a 0-100 mm visual analog scale.
P2 - Perceived risk of falling during daily ambulation with preferred assistive device/orthosis (Visual Analog Scale) | Baseline (single time point, within 24-month recruitment period)
  P2 assessed the patient's perceived risk of falling during daily ambulation with their preferred assistive device or orthosis on a 0-100 mm visual analog scale.
  Time Frame: Baseline (single time point, within 24-month recruitment period)
P3 - Perceived overall mobility compared to self-perceived maximum potential (Visual Analog Scale) | Baseline (single time point, within 24-month recruitment period)
  P3 assessed perceived overall mobility compared to the patient's self-perceived maximum potential on a 0-100 mm visual analog scale.
P4 - Degree of use of the most appropriate assistive device/orthosis during upright daily activities (Visual Analog Scale) | Baseline (single time point, within 24-month recruitment period)
  P4 assessed the degree to which the most appropriate assistive device or orthosis was used during upright daily activities on a 0-100 mm visual analog scale.
P5 - Comfort when using assistive devices/orthoses for walking or standing (Visual Analog Scale) | Baseline (single time point, within 24-month recruitment period)
  P5 assessed comfort when using assistive devices or orthoses for walking or standing on a 0-100 mm visual analog scale.
P6 - Perceived difficulty when using assistive devices/orthoses for walking or standing (Visual Analog Scale) | Baseline (single time point, within 24-month recruitment period)
  P6 assessed perceived difficulty when using assistive devices or orthoses for walking or standing on a 0-100 mm Visual Analog Scale.
P7 - Fatigue after using assistive devices/orthoses for 30-40 minutes in a single session (Visual Analog Scale) | Baseline (single time point, within 24-month recruitment period)
  P7 assessed fatigue experienced after using assistive devices or orthoses for 30-40 minutes in a single session on a 0-100 mm Visual Analog Scale.
P8 - Proportion of upright daily activities performed with walking aids (Visual Analog Scale) | Baseline (single time point, within 24-month recruitment period)
  P8 assessed the proportion of upright daily activities performed with walking aids on a 0-100 mm Visual Analog Scale.
P9 - Proportion of upright daily activities performed with seating aids (Visual Analog Scale) | Baseline (single time point, within 24-month recruitment period)
  P9 assessed the proportion of upright daily activities performed with seating aids such as wheelchairs on a 0-100 mm Visual Analog Scale.
P10 - Average daily hours spent standing (self-reported) | Baseline (single time point, within 24-month recruitment period)
  P10 recorded the average daily hours spent standing as reported by the patient.
P11 - Average daily hours spent sitting (self-reported) | Baseline (single time point, within 24-month recruitment period)
  P11 recorded the average daily hours spent sitting as reported by the patient.
P12 - Average daily hours spent lying down (self-reported) | Baseline (single time point, within 24-month recruitment period)
  P12 recorded the average daily hours spent lying down as reported by the patient.
P14 - Assistive device/orthosis planned for use in indoor ambulation after hospital discharge (Walking Index for Spinal Cord Injury II adapted categorical item) | Baseline (single time point, within 24-month recruitment period)
  P14 recorded the assistive device or orthosis planned for indoor ambulation after discharge, adapted from Walking Index for Spinal Cord Injury II categories.
P15 - Assistive device/orthosis planned for use in outdoor ambulation after hospital discharge (Walking Index for Spinal Cord Injury II adapted categorical item) | Baseline (single time point, within 24-month recruitment period)
  P15 recorded the assistive device or orthosis planned for outdoor ambulation after discharge, adapted from Walking Index for Spinal Cord Injury II categories.
P16 - Type of assistive device/orthosis used for outdoor ambulation over short distances during therapy (Walking Index for Spinal Cord Injury II adapted categorical item) | Baseline (single time point, within 24-month recruitment period)
  P16 recorded the type of assistive device or orthosis used for outdoor ambulation over short distances during therapy, adapted from Walking Index for Spinal Cord Injury II categories.
P17 - Number of falls within the past year in therapy and non-therapy settings (self-reported count) | Baseline (single time point, within 24-month recruitment period)
  P17 recorded the number of falls within the past year in therapy and non-therapy settings as self-reported by the patient.
P18 - Number of near-fall incidents within the past year in therapy and non-therapy settings (self-reported count) | Baseline (single time point, within 24-month recruitment period)
  P18 recorded the number of near-fall incidents within the past year in therapy and non-therapy settings as self-reported by the patient.
P19 - Assistive device/orthosis expected to be used in daily life after discharge (Walking Index for Spinal Cord Injury II adapted categorical item) | Baseline (single time point, within 24-month recruitment period)
  P19 recorded the assistive device or orthosis expected to be used in daily life after discharge, adapted from Walking Index for Spinal Cord Injury II categories.
T1 - Perceived patient's fall risk during daily ambulation with preferred assistive device/orthosis (Visual Analog Scale) | Baseline (single time point, within 24-month recruitment period)
  T1 assessed the therapist's perception of the patient's fall risk during daily ambulation with their preferred assistive device or orthosis on a 0-100 mm Visual Analog Scale.
T2 - Overall mobility compared to the patient's maximum potential (Visual Analog Scale) | Baseline (single time point, within 24-month recruitment period)
  T2 assessed the therapist's perception of the patient's overall mobility compared to their maximum potential on a 0-100 mm Visual Analog Scale.
T3 - Mobility level compared to a similar person without the injury (Visual Analog Scale) | Baseline (single time point, within 24-month recruitment period)
  T3 assessed the therapist's perception of the patient's mobility level compared to a similar person without injury on a 0-100 mm Visual Analog Scale.
T4 - Degree of use of the most appropriate assistive device/orthosis during upright daily activities without therapist guidance (Visual Analog Scale) | Baseline (single time point, within 24-month recruitment period)
  T4 assessed the degree to which the patient used the most appropriate assistive device or orthosis during upright daily activities without therapist guidance, on a 0-100 mm Visual Analog Scale.
T6 - Type of assistive device/orthosis used for outdoor ambulation over short distances during therapy (Walking Index for Spinal Cord Injury II adapted categorical item) | Baseline (single time point, within 24-month recruitment period)
  T6 recorded the type of assistive device or orthosis used for outdoor ambulation over short distances during therapy, adapted from Walking Index for Spinal Cord Injury II categories.
T7 - Assistive device/orthosis recommended for daily life after discharge (Walking Index for Spinal Cord Injury II adapted categorical item) | Baseline (single time point, within 24-month recruitment period)
  T7 recorded the assistive device or orthosis recommended for daily life after discharge, adapted from Walking Index for Spinal Cord Injury II categories.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Çankaya, Ankara, Turkey (Türkiye)